CLINICAL TRIAL: NCT05611619
Title: Low Particle Emission and Low Noise Tyres
Acronym: LEON-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: University of Pennsylvania (Other); University of Manitoba (Other); Swedish National Road and Transport Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 254066204
Record Dates: First submitted 2022-09-23; First posted 2022-11-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Noise Exposure; Sleep Disturbance; Sleep Hygiene; Metabolic Disturbance; Cognitive Change
Keywords: Neurobehavioural Performance; Polysomnography; Metabolomics
MeSH Terms: conditions — Parasomnias; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: There will be two separate study periods, each one affording the opportunity to investigate different acoustical characteristics of tyre noise and their physiological effects. Each of these study arms has a prospective within-subjects cross-over design. The order of the noise exposure conditions will be be randomly assigned across participants using a Latin square design to avoid first-order carryover effects. Each subject will be exposed to one night of each of the following:
  One quiet night: No noise will be played, serving as a control night to assess individual baseline sleep, cardiometabolic profile, and cognitive performance;
  Four traffic noise nights: Tyre noise from road traffic noise be played into the rooms to determine the effects of noise on sleep, cardiometabolic function and cognitive performance. These noise nights will be in a 2×2 factorial design so that we can examine each combination of two specific noise characteristics.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be aware that in any given study night they can be exposed to traffic noise. They will not be informed what noise condition will occur in any given night, but they can become unblinded to the exposure if they are awake, as they will hear the noise.
  Study investigators responsible for analysing cognitive performance variables and physiological sleep data will be be blind to which noise interventions were introduced on which study nights.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Control (No Intervention): Single study night with no noise exposure, to determine normal baseline sleep
- Study 1: High level continuous flow tyre noise (A1) (Experimental): Single study night in first experimental study arm, with traffic noise to determine consequences of sleep disturbance by high level, continuous flow traffic noise. Noise will include mix of different acoustical characteristics of tyre noise throughout the night.
  Interventions: Radiation: Tyre noise - continuous flow; Radiation: High noise level
- Study 1: Medium level continuous flow tyre noise (B1) (Experimental): Single study night in first experimental study arm, with traffic noise to determine consequences of sleep disturbance by medium level, continuous flow traffic noise. Noise will include mix of different acoustical characteristics of tyre noise throughout the night.
  Interventions: Radiation: Tyre noise - continuous flow; Radiation: Moderate noise level
- Study 1: High level, discrete traffic tyre noise (A2) (Experimental): Single study night in first experimental study arm, with traffic noise events to determine consequences of sleep disturbance by high level traffic noise comprised of single, discrete traffic events. Noise will include mix of different acoustical characteristics of tyre noise throughout the night.
  Interventions: Radiation: Tyre noise - discrete events; Radiation: High noise level
- Study 1: Medium level, discrete traffic tyre noise (B2) (Experimental): Single study night in first experimental study arm, with traffic noise events to determine consequences of sleep disturbance by moderate level traffic noise comprised of single, discrete traffic events. Noise will include mix of different acoustical characteristics of tyre noise throughout the night.
  Interventions: Radiation: Tyre noise - discrete events; Radiation: Moderate noise level
- Study 2: Medium level composite wheel tyre noise (A1) (Experimental): Single study night in second experimental study arm, with traffic noise to determine consequences of sleep disturbance by medium level traffic noise comprised of composite wheel types.
  Interventions: Radiation: Moderate noise level; Radiation: Composite tyres
- Study 2: Low level composite wheel tyre noise (B1) (Experimental): Single study night in second experimental study arm, with traffic noise to determine consequences of sleep disturbance by low level traffic noise comprised of composite wheel types.
  Interventions: Radiation: Low noise level; Radiation: Composite tyres
- Study 2: Medium level air-filled tyre noise (A2) (Experimental): Single study night in second experimental study arm, with traffic noise to determine consequences of sleep disturbance by medium level traffic noise comprised of traditional air-filled wheel types.
  Interventions: Radiation: Moderate noise level; Radiation: Air-filled tyres
- Study 2: Low level air-filled tyre noise (B2) (Experimental): Single study night in second experimental study arm, with traffic noise to determine consequences of sleep disturbance by low level traffic noise comprised of traditional air-filled wheel types.
  Interventions: Radiation: Low noise level; Radiation: Air-filled tyres

INTERVENTIONS:
Radiation: Tyre noise - continuous flow — Tyre noise from continuous traffic, throughout the night
  Arms: Study 1: High level continuous flow tyre noise (A1); Study 1: Medium level continuous flow tyre noise (B1)
Radiation: Tyre noise - discrete events — Tyre noise from few, discrete traffic events, occurring throughout the night
  Arms: Study 1: High level, discrete traffic tyre noise (A2); Study 1: Medium level, discrete traffic tyre noise (B2)
Radiation: High noise level — Tyre noise corresponding up to 65 dB LAEq,24h
  Arms: Study 1: High level continuous flow tyre noise (A1); Study 1: High level, discrete traffic tyre noise (A2)
Radiation: Moderate noise level — Tyre noise corresponding up to 60 dB LAEq,24h
  Arms: Study 1: Medium level continuous flow tyre noise (B1); Study 1: Medium level, discrete traffic tyre noise (B2); Study 2: Medium level air-filled tyre noise (A2); Study 2: Medium level composite wheel tyre noise (A1)
Radiation: Low noise level — Tyre noise corresponding up to 55 dB LAEq,24h
  Arms: Study 2: Low level air-filled tyre noise (B2); Study 2: Low level composite wheel tyre noise (B1)
Radiation: Air-filled tyres — Tyre noise from traditional, air-filled tyres
  Arms: Study 2: Low level air-filled tyre noise (B2); Study 2: Medium level air-filled tyre noise (A2)
Radiation: Composite tyres — Tyre noise from newly designed, airless composite tyres
  Arms: Study 2: Low level composite wheel tyre noise (B1); Study 2: Medium level composite wheel tyre noise (A1)

SUMMARY:
This study will investigate the biological mechanisms linking sleep disruption by noise and the development of disease. In a laboratory sleep study, the investigators will play synthesised automotive tyre sounds, investigating how acoustical characteristics of tyre noise impact on sleep macrostructure, cardiometabolic profile and cognitive performance (continuous traffic flow or a few individual, but higher level, traffic pass-bys). The investigators will also measure objective sleep quality and quantity, cognitive performance across multiple domains, self-reported sleep and wellbeing outcomes, and blood samples. Blood samples will be analysed to identify metabolic changes in different nights. Identifying biomarkers that are impacted by sleep fragmentation will establish the currently unclear pathways by which chronic noise exposure at night can lead to the development of diseases in the long term, especially cardiometabolic disorders.

DETAILED DESCRIPTION:
The experimental sleep study has the overarching goal of deepening our understanding of sleep disruption by automotive tyre noise and changes in cardiometabolic and cognitive function. To this end, the study will address the following independent aims:

Aim 1: Determine the biological and neurobehavioural consequences of sleep disruption by tyre noise. The investigators will measure the sleep of healthy volunteers, and each morning the investigators will obtain blood samples for metabolomics analysis and administer a neurocognitive test battery. The investigators will compare effects on sleep, metabolomics and cognitive function between quiet nights and nights with road traffic noise.

Aim 2: Identify acoustical characteristics of tyre noise that are especially disturbing physiologically. The investigators will use different combinations of types of tyre noise in different noise exposure nights to determine differential effects on sleep and cardiovascular response.

This study will take place in the sound environment laboratory (SEL) at the University of Gothenburg Department of Occupational and Environmental Medicine (Arbets- och miljömedicin [AMM]). The SEL is a high fidelity research laboratory equipped to simulate a typical apartment, including three individually light-, sound- and vibration-isolated private bedrooms. Ceiling mounted speakers in each room allow the investigators to create a realistic acoustic environment by transmitting sound exposures from the control room to each bedroom individually. The investigators have shown previously that results from this lab with high ecological validity are comparable with results from the field.

There will be two study arms, each one affording the opportunity to investigate different acoustical characteristics of tyre noise and their physiological effects. Each of these study arms has a prospective within-subjects cross-over design. Participants (study 1 N=15; study 2 N=30; total N=45 across both arms) will each spend six consecutive nights in the SEL, with a sleep opportunity between 23:00-07:00. Daytime sleep will be prohibited, confirmed with measures of daytime activity via wrist actigraphy monitors worn continuously throughout the study. Three subjects will take part concurrently, in separate bedrooms. The first night is a habituation period to the study protocol and for familiarisation with the test procedures. Study nights 2-6 are the experimental nights and will be randomly assigned across participants using a Latin square design to avoid first-order carryover effects. Each subject will be exposed to each of the following:

One quiet night: No noise will be played, serving as a control night to assess individual baseline sleep, cardiometabolic profile, and cognitive performance;

Four traffic noise nights: Tyre noise from road traffic noise be played into the rooms to determine the effects of noise on sleep, cardiometabolic function and cognitive performance. These noise nights will be in a 2×2 factorial design so that the investigators can examine each combination of two specific noise characteristics.

Each night the investigators will record physiologic sleep with polysomnography (PSG) and cardiac activity with electrocardiography (ECG). Each study morning, subjects will provide a 4 ml blood sample, complete cognitive testing and answer questionnaires and will depart the SEL to follow their normal daytime routine. They will return to the SEL at 20:00 each evening to prepare for sleep measurements. Caffeine will be prohibited after 15:00 and alcohol will be prohibited at all times. Because extreme and/or variable dietary behaviour can affect the metabolome/lipoprotein profile, participants will be given guidance that they should eat a similar evening meal on each day of the laboratory study, confirmed with a food diary, The actual meal itself can be different for different study participants, because the study has a within-subjects design.

Sleep will be recorded with ambulatory polysomnography (PSG) and cardiac activity with electrocardiography (ECG) and finger pulse photoplethysmogram. Data are recorded offline onto the sleep recorder, and will be downloaded and checked every study morning to ensure data quality. In addition to traditional sleep analysis performed by the research group at the University of Gothenburg, raw PSG data will be used to calculate the Odds Ratio Project, a novel metric of sleep depth and stability.

Each study morning subjects will provide a 4 ml blood sample for plasma metabolomics analysis. To ensure reliable data, blood samples will be taken at the same time every day to mitigate circadian effects, before eating or drinking anything except water, and each sample will be handled in the same way i.e. centrifuged, aliquoted and stored in -80C freezers. Subjects will eat the same food each study evening to mitigate within-subject dietary effects on the blood metabolome.

Each morning, subjects will complete a computerised cognitive test battery taking approximately 20 minutes, that includes 10 tests across a range of cognitive domains (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance). Cognition data will be analysed to determine key measures of cognitive speed and accuracy, adjusting for practice effects and the difficulty of the stimulus set.

Subjects will complete a battery of one-time validated questionnaires to measure their general health (SF-36), chronotype, noise sensitivity, habitual sleep quality, environmental sensitivity, and annoyance and sleep disturbance by noise. Subjects will also answer a questionnaire each study evening and morning, involving questions on sleepiness (Karolinska Sleepiness Scale), sleep disturbance by noise, positive and negative affect (PANAS), and validated sleep and disturbance questions.

Participants will wear a wrist actigraphy monitor continuously throughout the study period, and also for the week before the study, to confirm habitual sleep-wake times and to measure physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

1. live in or around the city of Gothenburg area (Sweden)

Exclusion Criteria:

1. aged <18 or >30 years;
2. habitual sleep and wake timings more than ±1 hour different from the study sleep times (i.e. habitual sleep time should be 22:00-00:00 and habitual wake time should be 06:00-08:00);
3. BMI>25 kg/m2;
4. regular sleep medication use (prescribed or "over-the-counter");
5. poor hearing acuity (measured during screening via pure tone audiometry);
6. diagnosed with sleep disorders;
7. indications of sleep apnea on the STOP-BANG questionnaire;
8. shift work;
9. smoking, vaping, snus, or other nicotine use.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Baseline total sleep time during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline total sleep time during the A1 night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline total sleep time during the A2 night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline total sleep time during the B1 night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline total sleep time during the B2 night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during exposure to nocturnal tyre noise combination A1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during exposure to nocturnal tyre noise combination A2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during exposure to nocturnal tyre noise combination B1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total sleep time during exposure to nocturnal tyre noise combination B2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline N1 sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline N2 sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline N3 sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of baseline rapid eye movement (REM) sleep during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during exposure to nocturnal tyre noise combination A1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during exposure to nocturnal tyre noise combination A1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during exposure to nocturnal tyre noise combination A1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during exposure to nocturnal tyre noise combination A1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during exposure to nocturnal tyre noise combination A2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during exposure to nocturnal tyre noise combination A2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during exposure to nocturnal tyre noise combination A2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during exposure to nocturnal tyre noise combination A2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during exposure to nocturnal tyre noise combination B1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during exposure to nocturnal tyre noise combination B1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during exposure to nocturnal tyre noise combination B1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during exposure to nocturnal tyre noise combination B1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N1 sleep during exposure to nocturnal tyre noise combination B2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N2 sleep during exposure to nocturnal tyre noise combination B2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of N3 sleep during exposure to nocturnal tyre noise combination B2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Total amount of rapid eye movement (REM) sleep during exposure to nocturnal tyre noise combination B2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline wakefulness after sleep onset (WASO) during the Control night | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during exposure to nocturnal tyre noise combination A1 | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during exposure to nocturnal tyre noise combination A2 | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during exposure to nocturnal tyre noise combination B1 | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Wakefulness after sleep onset (WASO) during exposure to nocturnal tyre noise combination B2 | One night
  Total number of minutes awake during the night after the first appearance of sleep of any stage. Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline number of awakenings during the Control night | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Number of awakenings during exposure to nocturnal tyre noise combination A1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Number of awakenings during exposure to nocturnal tyre noise combination A2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Number of awakenings during exposure to nocturnal tyre noise combination B1 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Number of awakenings during exposure to nocturnal tyre noise combination B2 | One night
  Measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines
Baseline sleep onset latency (SOL) during the Control night | One night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during exposure to nocturnal tyre noise combination A1 | One night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during exposure to nocturnal tyre noise combination A2 | One night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during exposure to nocturnal tyre noise combination B1 | One night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep onset latency (SOL) during exposure to nocturnal tyre noise combination B2 | One night
  Defined as the time from lights out to the first epoch of sleep measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Baseline sleep efficiency during the Control night | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during exposure to nocturnal tyre noise combination A1 | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during exposure to nocturnal tyre noise combination A2 | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during exposure to nocturnal tyre noise combination B1 | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Sleep efficiency during exposure to nocturnal tyre noise combination B2 | One night
  Defined as the percentage of time in bed spent in a non-wake sleep stage, measured via polysomnography/EEG, scored according to American Academy of Sleep Medicine guidelines.
Baseline sleep depth assessed using the odds ratio product (ORP) during the Control night | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during exposure to nocturnal tyre noise combination A1 | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during exposure to nocturnal tyre noise combination A2 | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during exposure to nocturnal tyre noise combination B1 | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Sleep depth assessed using the odds ratio product (ORP) during exposure to nocturnal tyre noise combination B2 | One night
  Average ORP over the full night, from 0 (never occurs during wake) to 2.5 (only occurs during wake). Derived via polysomnography/EEG measurements.
Spontaneous maximal change of odds ratio product (ORP) during the Control night | One night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over 120 sham noise events during the night.
Maximal change of odds ratio product (ORP) during exposure to tyre noise events combination A1 | One night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over all 120 noise events during the night.
Maximal change of odds ratio product (ORP) during exposure to tyre noise events combination A2 | One night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over all 120 noise events during the night.
Maximal change of odds ratio product (ORP) during exposure to tyre noise events combination B1 | One night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over all 120 noise events during the night.
Maximal change of odds ratio product (ORP) during exposure to tyre noise events combination B2 | One night
  Primary measure of acute sleep disruption by noise, calculated as the difference between the ORP in the 30s prior to noise onset and the maximum ORP during traffic noise. Averaged over all 120 noise events during the night.
Morning neurobehavioural speed in the morning immediately after the Control night | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural speed in the morning immediately after the A1 night | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural speed in the morning immediately after the A2 night | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural speed in the morning immediately after the B1 night | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural speed in the morning immediately after the B2 night | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Morning neurobehavioural accuracy in the morning after the control night | One night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Morning neurobehavioural accuracy in the morning after exposure to nocturnal tyre noise combination A1 | One night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Morning neurobehavioural accuracy in the morning after exposure to nocturnal tyre noise combination A2 | One night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Morning neurobehavioural accuracy in the morning after exposure to nocturnal tyre noise combination B1 | One night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Morning neurobehavioural accuracy in the morning after exposure to nocturnal tyre noise combination B2 | One night
  Average of one key accuracy indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Baseline evening neurobehavioural speed following the Control night | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural speed after exposure to nocturnal tyre noise combination A1 | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural speed after exposure to nocturnal tyre noise combination A2 | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural speed after exposure to nocturnal tyre noise combination B1 | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Evening neurobehavioural speed after exposure to nocturnal tyre noise combination B2 | One night
  Average of one key speed indicator from each of 10 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, balloon analog risk, psychomotor vigilance)
Baseline evening neurobehavioural accuracy following the Control night | One night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance
Evening neurobehavioural accuracy after exposure to nocturnal tyre noise combination A1 | One night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Evening neurobehavioural accuracy after exposure to nocturnal tyre noise combination A2 | One night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Evening neurobehavioural accuracy after exposure to nocturnal tyre noise combination B1 | One night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Evening neurobehavioural accuracy after exposure to nocturnal tyre noise combination B2 | One night
  Average of one key speed indicator from each of 9 cognitive tests (motor praxis, visual object learning, fractal 2-back, abstract matching, line orientation, emotion recognition, matrix reasoning, digit symbol substitution, psychomotor vigilance)
Event-related Cardiovascular activation in response to noise during Control night | One night
  Change in heart rate (ECG)
Event-related Cardiovascular activation in response to noise during A1 | One night
  Change in heart rate (ECG)
Event-related Cardiovascular activation in response to noise during A2 | One night
  Change in heart rate (ECG)
Event-related Cardiovascular activation in response to noise during B1 | One night
  Change in heart rate (ECG)
Event-related Cardiovascular activation in response to noise during B2 | One night
  Change in heart rate (ECG)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale on the control night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale on the A1 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale on the A2 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale on the B1 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Evening subjective sleepiness, assessed using the Karolinska Sleepiness Scale on the B2 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after the control night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after the A1 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after the A2 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after the B1 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Morning subjective sleepiness, assessed using the Karolinska Sleepiness Scale after the B2 night | One night
  The scale is a 9-level verbal scale from 1 - "Extremely alert" (best outcome) to 9 - "Very sleepy. great effort to keep alert, fighting sleep" (worst outcome)
Taurine concentration (mmol/L) immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Taurine concentration (mmol/L) in the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Taurine concentration (mmol/L) in the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Taurine concentration (mmol/L) in the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Taurine concentration (mmol/L) in the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Serotonin concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Serotonin concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Serotonin concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Serotonin concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Serotonin concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Tryptophan concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Tryptophan concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Tryptophan concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Tryptophan concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Tryptophan concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Isoleucine concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Isoleucine concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Isoleucine concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Isoleucine concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Isoleucine concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Leucine concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Leucine concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Leucine concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Leucine concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Leucine concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Valine concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Valine concentration (mmol/L)In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Valine concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Valine concentration (mmol/L)In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Valine concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Diacylglycerol (36:3) concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Diacylglycerol (36:3) concentration (mmol/L)In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Diacylglycerol (36:3) concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Diacylglycerol (36:3) concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Diacylglycerol (36:3) concentration (mmol/L)In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Lauroylcarnitine (C12:0) concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Lauroylcarnitine (C12:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Lauroylcarnitine (C12:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Lauroylcarnitine (C12:0) concentration (mmol/L)In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Lauroylcarnitine (C12:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Octanoylcarnitine (C8:0) concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Octanoylcarnitine (C8:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Octanoylcarnitine (C8:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Octanoylcarnitine (C8:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Octanoylcarnitine (C8:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Myristoylcarnitine (C14:0) concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Myristoylcarnitine (C14:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Myristoylcarnitine (C14:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Myristoylcarnitine (C14:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Myristoylcarnitine (C14:0) concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline 1-Methyl-4-pyridone-5-carboxamide (4-Pyr) concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
1-Methyl-4-pyridone-5-carboxamide (4-Pyr) concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
1-Methyl-4-pyridone-5-carboxamide (4-Pyr) concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
1-Methyl-4-pyridone-5-carboxamide (4-Pyr) concentration (mmol/L)In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
1-Methyl-4-pyridone-5-carboxamide (4-Pyr) concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Phenylalanine concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Phenylalanine concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Phenylalanine concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Phenylalanine concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Phenylalanine concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Acylcarnitine C18:1 concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C18:1 concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C18:1 concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C18:1 concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C18:1 concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Acylcarnitine C10:0 concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C10:0 concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C10:0 concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C10:0 concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Acylcarnitine C10:0 concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Phosphatidylcholine 32:1 concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 32:1 concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 32:1 concentration (mmol/L)In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 32:1 concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 32:1 concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Basline Phosphatidylcholine 38:2 concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:2 concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:2 concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:2 concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:2 concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma
Baseline Phosphatidylcholine 38:3 concentration (mmol/L) In the morning immediately after the Control night | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:3 concentration (mmol/L) In the morning immediately after the Tyre noise combination A1 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:3 concentration (mmol/L) In the morning immediately after the Tyre noise combination A2 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:3 concentration (mmol/L) In the morning immediately after the Tyre noise combination B1 | One night
  Determined from GC-MS analysis of blood plasma
Phosphatidylcholine 38:3 concentration (mmol/L) In the morning immediately after the Tyre noise combination B2 | One night
  Determined from GC-MS analysis of blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Smith, PhD, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No